CLINICAL TRIAL: NCT05393102
Title: Auxiliary Diagnosis of Liver Nodules Using cfDNA Whole-genome SignatuRes (GUDIER): an Observational Cohort Trial
Brief Title: Auxiliary Diagnosis of Liver Nodules Using cfDNA Whole-genome Signatures
Acronym: GUIDER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Hong Ren, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2022-20
Record Dates: First submitted 2022-05-08; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Focal Liver Lesions
Keywords: hepatocellular carcinoma; liver nodules; auxiliary diagnosis; liquid biopsy; peripheral blood; cfDNA
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Malignant liver nodules cohort: Participants with malignant liver nodules diagnosed by pathological biopsy.
  Interventions: Other: No interventions
- Benign liver nodules cohort: Participants with benign liver nodules diagnosed by pathological biopsy or imaging examination.
  Interventions: Other: No interventions
- Uncertain benign or malignant liver nodules cohort: Participants with liver nodules could not be diagnosed definitely by imaging examination and serum protein markers.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions

SUMMARY:
As a prospective, multi-center study, GUIDER will recruit 400 liver nodules participants from different provinces and regions across China. Except for cfDNA signatures, serum biomarkers, histopathological biopsy and enhanced MRI will also be performed. The sensitivity and specificity of the cfDNA signature based-model in liver nodules diagnosing will be evaluated.

DETAILED DESCRIPTION:
Patients with liver nodules will be recruited for 1 year. Peripheral blood samples of all participants will be collected after being informed about the study and potential risks. CfDNA extraction, library construction, and whole genome sequencing will be performed. A machine learning method will be implemented for cfDNA signatures-based model construction at the end of the study. Sensitivity and specificity will be used to evaluate the performance of cfDNA signatures-based model in liver nodules diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years or elder；
* Participants underwent enhanced MRI for the evaluation of liver nodules ≤5 cm；
* Participants whose platelet count ≥ 50×109/L, prothrombin activity (PTA) ≥ 60%；
* Participants who are willing and able to perform hepatectomy or tissure biopsy.

Exclusion Criteria:

* Participants with different enhancement mode liver nodules that detected by enhanced MRI and without CEUS confirmation；
* Diagnosis of malignant tumors before recruitment；
* Anti-tumor therapy before recruitment ；
* HIV infection；
* Pregnancy；
* Allogenic blood transfusion or cell therapy within 14 days before peripheral blood samples collection;
* Participants with hepatic encephalopathy, hemangioma, ascites, gastrointestinal bleeding, jaundice, liver failure, congestive heart failure, or any other serious diseases that causing organ damage.
* Participants with any other factors that may leading to termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Four hundreds eligible participants will be recruited from medical centers and assigned into three groups, including participants with malignant or benign liver nodules，and participants with uncertain liver nodules.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the cfDNA whole-genome signatures based model in liver nodules diagnosis. | Enrollment of the first participant up to 18 months
  Sensitivity is defined as the ratio of positively detected participants in all malignant nodule patients by cfDNA signatures.
Specificity of the cfDNA whole-genome signatures based model in liver nodules diagnosis. | Enrollment of the first participant up to 18 months
  Specificity is defined as the proportion of negatively detected participants in all benign liver nodules patients by cfDNA signatures.

SECONDARY OUTCOMES:
Specificity of the model that composed of cfDNA signatures, imaging examination，serum protein markers and clinical characteristics in liver nodules diagnosis. | Through study completion，an average of 18 months
  Specificity is defined as the proportion of negatively detected participants in all benign liver nodules patients by the model that composed of cfDNA whole-genome signatures, imaging examination，serum protein markers， and clinical characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, MD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University; Hongyang Wang, MD, Principal Investigator — Eastern Hepatobiliary Surgery Hospita; Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (3):
- China (3):
  - The 2nd affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Kobayashi M, Ikeda K, Hosaka T, Sezaki H, Someya T, Akuta N, Suzuki F, Suzuki Y, Saitoh S, Arase Y, Kumada H. Dysplastic nodules frequently develop into hepatocellular carcinoma in patients with chronic viral hepatitis and cirrhosis. Cancer. 2006 Feb 1;106(3):636-47. doi: 10.1002/cncr.21607. PMID 16369988
- [Background] Llovet JM, Chen Y, Wurmbach E, Roayaie S, Fiel MI, Schwartz M, Thung SN, Khitrov G, Zhang W, Villanueva A, Battiston C, Mazzaferro V, Bruix J, Waxman S, Friedman SL. A molecular signature to discriminate dysplastic nodules from early hepatocellular carcinoma in HCV cirrhosis. Gastroenterology. 2006 Dec;131(6):1758-67. doi: 10.1053/j.gastro.2006.09.014. Epub 2006 Sep 19. PMID 17087938
- [Background] Chen L, Abou-Alfa GK, Zheng B, Liu JF, Bai J, Du LT, Qian YS, Fan R, Liu XL, Wu L, Hou JL, Wang HY; PreCar Team. Genome-scale profiling of circulating cell-free DNA signatures for early detection of hepatocellular carcinoma in cirrhotic patients. Cell Res. 2021 May;31(5):589-592. doi: 10.1038/s41422-020-00457-7. Epub 2021 Feb 15. No abstract available. PMID 33589745